CLINICAL TRIAL: NCT04246034
Title: Evaluation of Outcomes of Microvascular Breast Reconstruction With Lymph Node Transfer for Postmastectomy Lymphedema Patients
Brief Title: Microvascular Breast Reconstruction With Lymph Node Transfer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: surgery considered elective and cant be performed within corona restrictions
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed ElSayed Sharaf Ahmed, Assistant Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VLNT for lymphedema
Record Dates: First submitted 2020-01-18; First posted 2020-01-29 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Lymphedema; Lymphedema of Upper Arm; Mastectomy; Lymphedema
Keywords: VLNT; breast reconstruction; postmastectomy lymphedema; vascularized lymph node transfer; lymphedema surgery; microsurgery
MeSH Terms: conditions — Lymphedema; Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cases (Experimental): As described by Saaristo et al. in 2012, the surgical technique starts with wide axillary scar removal, followed by elevation of contralateral dual flap which includes DIEP/MS-TRAM with attached groin lymph nodes and fat, then the anastomosis is preferably done to internal mammary vessels.
  Interventions: Procedure: Microvascular Breast Reconstruction with Vascularized Lymph Node Transfer

INTERVENTIONS:
Procedure: Microvascular Breast Reconstruction with Vascularized Lymph Node Transfer — simultaneous free abdominal flaps with VLNT from groin are transferred on a single pedicle for breast reconstruction and postmastectomy lymphedema

SUMMARY:
this study aims to evaluate the outcomes of simultaneous free abdominal flap & vascularized lymph node transfer for both breast reconstruction and postmastectomy lymphedema

DETAILED DESCRIPTION:
Microvascular breast reconstruction allows for the transfer of donor tissue that is an excellent match for native breast tissue, both in terms of the subcutaneous tissue that reconstitutes the breast mound and the simultaneous transfer of skin. In addition, it offers a wide range of options for women who may have been previously not considered for autologous tissue transfer. From the these various options, the deep inferior epigastric artery perforator (DIEP) flap and the muscle-sparing transverse rectus abdominis myocutaneous (MS-TRAM) flap are the most recognized free flap options for breast reconstruction today

Besides the needs for breast reconstruction after mastectomy & axillary lymph node dissection, upper limb lymphedema is also a major concern for postmastectomy patients which is estimated to occur in 21.4% of women treated for breast cancer. It represents a diagnostic and therapeutic challenge for clinicians due to the heterogeneity in presentation as well as multitude of treatment options available. In addition, with a lack of evidence-based guidelines

. According to the International Society of Lymphology Consensus, the clinical staging of lymphedema includes; Stage 0 (Subclinical) when lymphatic vessels have been injured but have no measurable swelling or edema. Stage I lymphedema occurs with the onset of measurable swelling and pitting of the skin which can be regressed on conservative treatments. Stage II considered when there is edema partially regressing with treatments and negative pitting test. Stage III encompasses lymphostatic elephantiasis with trophic skin changes and recurrent infections.

In recent years, lymphatic microsurgery procedures have increased in popularity, bringing in a new wave of physiologic surgical options for the management of lymphedema. The two most common microsurgical options include lymphovenous anastomosis (LVA) and vascularized lymph node transfer (VLNT). Each treatment option has the potential to bypass areas of damaged lymphatics by rerouting the lymph into the venous system or by replacing the lost lymph nodes and, or lymphatic ducts.

Recent studies have evaluated the positive effects of VLNT in the setting of lymphedema and have shown significantly better results for the patients in which the native lymphatic ducts are no longer available when compared to conservative treatments or LVA.

There are several potential donor sites that can be used for the VLNT, and currently, there is no clear consensus as to which lymph node basin represents the ideal donor site. But the most popular lymph nodes have been the supraclavicular nodes, the submental nodes, the lateral thoracic nodes, the inguinal nodes, the omentum, and more recently the mesenteric lymph nodes. However, in patients suffering from post-mastectomy lymphedema, the inguinal nodes can be transferred at the time of autologous breast reconstruction, coupling the inguinal nodes to (DIEP) flap or (MS-TRAM) flap to reconstruct the patient's breast while simultaneously addressing the patient's lymphedema in one operation .

Advantages of simultaneous breast reconstruction & VLNT include the extensive scar removal and release in the axilla, which is critical to optimizing the recipient bed for the VLNT and the relatively hidden scar in axilla. Although a promising technique, it remains investigational and requires larger studies with longer follow-up to validate its true utility. Of primary concern is monitoring for the longevity of the results and making certain that additional donor site morbidity is avoided.

To the best of the investigator's knowledge, few studies were conducted on the use of free abdominal free flaps in conjunction with VLNT from the groin for simultaneous lymphedema treatment & breast reconstruction. But these studies were limited by small sample sizes.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of 20-65 years old
* Patients seeking autologous breast reconstruction and complain of clinically diagnosed arm lymphedema
* Deficient lymphatic drainage on lymphoscintigraphy
* Stage II and III Lymphedema
* no active cellulitis
* more than 12 months of follow-up

Exclusion Criteria:

* Females < 20 or >65 years old
* distant metastasis
* brachial plexus neuritis.
* Patients with unhealthy and obstructed recipient veins or congestive heart disease with limited venous return may not be a suitable candidate for the procedure.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — as the scope of study is breast cancer, participant should be of female gender
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in upper limb volume | 6-12 months
  Assessment of volume reduction by measuring limb circumference of affected and non affected upper limbs at fixed points from shoulder, elbow & wrist joints
Change in lymphatic flow | 6-12 months
  lymphoscintigraphy will be used to trace radiological signs of Lymphatic flow improvement such as reduced dermal backflow, appearance of new lymph drainage channels, reduced stasis and increased rate of radiolabeled tracer clearance

SECONDARY OUTCOMES:
Quality of life measure for limb lymphedema (LYMQOL) | 6-12 months
  Quality of life parameters will be measured using LYMQOL survey. Questions in the survey cover four areas: symptoms, body image/appearance, function and mood. Answers are scored 1-4 (less severe to severe)
Quality of life measure for breast | 6-12 months
  patient quality of life will be evaluated using Breast-Q "Reconstruction Module", which includes different modules for assessment of quality of life and patient satisfaction after breast reconstruction. These scales are designed to be administered pre-operatively and assess patient expectations for the process and outcome of surgery. The expectations scales compliment the satisfaction and quality-of life domains of the postoperative reconstruction module. Multi-item and categorical scale structures are used. Five scales provide a 0-100 score. A higher score means better quality of life and more satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Youssef S Hassan, MD, Study Chair — Assiut University Hospitals - Plastic Surgery Dept.; Haitham Khalil, MD, FRCS, Study Director — Divison of Plastic and Reconstructive Surgery (University Hospitals Birmingham); Awny M Asklany, MD, Study Director — Assiut University Hospitals - Plastic Surgery Dept.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saaristo AM, Niemi TS, Viitanen TP, Tervala TV, Hartiala P, Suominen EA. Microvascular breast reconstruction and lymph node transfer for postmastectomy lymphedema patients. Ann Surg. 2012 Mar;255(3):468-73. doi: 10.1097/SLA.0b013e3182426757. PMID 22233832
- [Background] DiSipio T, Rye S, Newman B, Hayes S. Incidence of unilateral arm lymphoedema after breast cancer: a systematic review and meta-analysis. Lancet Oncol. 2013 May;14(6):500-15. doi: 10.1016/S1470-2045(13)70076-7. Epub 2013 Mar 27. PMID 23540561
- [Background] Smile TD, Tendulkar R, Schwarz G, Arthur D, Grobmyer S, Valente S, Vicini F, Shah C. A Review of Treatment for Breast Cancer-Related Lymphedema: Paradigms for Clinical Practice. Am J Clin Oncol. 2018 Feb;41(2):178-190. doi: 10.1097/COC.0000000000000355. PMID 28009597
- [Background] Executive Committee. The Diagnosis and Treatment of Peripheral Lymphedema: 2016 Consensus Document of the International Society of Lymphology. Lymphology. 2016 Dec;49(4):170-84. PMID 29908550
- [Background] Pappalardo M, Patel K, Cheng MH. Vascularized lymph node transfer for treatment of extremity lymphedema: An overview of current controversies regarding donor sites, recipient sites and outcomes. J Surg Oncol. 2018 Jun;117(7):1420-1431. doi: 10.1002/jso.25034. Epub 2018 Mar 24. PMID 29572824
- [Background] Engel H, Lin CY, Huang JJ, Cheng MH. Outcomes of Lymphedema Microsurgery for Breast Cancer-related Lymphedema With or Without Microvascular Breast Reconstruction. Ann Surg. 2018 Dec;268(6):1076-1083. doi: 10.1097/SLA.0000000000002322. PMID 28594742
- [Background] Chang EI, Masia J, Smith ML. Combining Autologous Breast Reconstruction and Vascularized Lymph Node Transfer. Semin Plast Surg. 2018 Feb;32(1):36-41. doi: 10.1055/s-0038-1632402. Epub 2018 Apr 9. PMID 29636652
- [Background] Nguyen AT, Chang EI, Suami H, Chang DW. An algorithmic approach to simultaneous vascularized lymph node transfer with microvascular breast reconstruction. Ann Surg Oncol. 2015 Sep;22(9):2919-24. doi: 10.1245/s10434-015-4408-4. Epub 2015 Jan 27. PMID 25623599